CLINICAL TRIAL: NCT07246291
Title: Randomized, Double-Blind, Parallel-Controlled, Single-Dose Pharmacokinetic, Safety, and Immunogenicity Comparative Study of EnliTuo® Before and After Technology Change in Healthy Male Volunteers
Brief Title: Comparative Study of EnliTuo® Before and After Technology Change in Healthy Male Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMAB009-C-102
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adult Male
Keywords: phrase 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New technology Enlituo (Experimental): treated with new technology Enlituo through single intravenous drip
  Interventions: Biological: New technology Enlituo
- Approved technology Enlituo (Active Comparator): treated with Approved technology Enlituo through single intravenous drip
  Interventions: Biological: Approved technology Enlituo

INTERVENTIONS:
Biological: New technology Enlituo — 250 mg/m^2, single intravenous drip
  Arms: New technology Enlituo
Biological: Approved technology Enlituo — 250 mg/m^2, single intravenous drip
  Arms: Approved technology Enlituo

SUMMARY:
This study is a randomized, double-Blind, parallel-controlled, single-dose pharmacokinetic, safety, and immunogenicity comparative study of EnliTuo® before and after technology change in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged ≥ 18 years and ≤ 45 years on the day of signing the informed consent form;
* At screening, body weight ≥ 50 kg and ≤ 80 kg, with a Body Mass Index (BMI) between 19.0 and 26.0 kg/m² (inclusive of boundary values);
* Capable of understanding the study, including its purpose, research procedures, potential risks, etc., and able to communicate well with researchers and complete the study in accordance with the study requirements;
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Subjects with any abnormally clinically significant findings in comprehensive examinations (vital signs, physical examination, electrocardiogram, chest X-ray, abdominal ultrasound, blood routine, urine routine, blood biochemistry, coagulation, etc.) as judged by the investigator;
* Subjects with a history of major diseases in the cardiovascular, endocrine, nervous, digestive, respiratory, genitourinary, hematological, immune, or mental systems, or currently suffering from any disease in the above systems;
* Subjects with a known or suspected history of keratitis, ulcerative keratitis, conjunctivitis, blepharitis, or severe dry eye;
* Subjects with hereditary bleeding tendency, coagulation dysfunction, or a history of thrombotic or hemorrhagic diseases;
* Subjects with active infections requiring systemic treatment;
* Subjects positive for any of HBV surface antigen, HCV antibody, HIV antibody, or Treponema pallidum antibody;
* Subjects with a history of malignant tumors within the past 5 years, except for completely resected in-situ cutaneous basal cell carcinoma or squamous cell carcinoma;
* Subjects who have undergone surgical operations within 4 weeks before screening, or plan to undergo surgery during the trial period;
* Subjects who have used any prescription drugs, over-the-counter drugs, traditional Chinese medicines, proprietary Chinese medicines, health supplements, etc., within 4 weeks before screening, or whose use of the above substances has not exceeded 5 half-lives (whichever is longer);
* Subjects who have used any biological products or received any vaccines within 12 weeks before screening, or plan to receive any vaccines during the study period;
* Subjects currently enrolled in other clinical studies of drugs or medical devices, or whose time since the end of the last enrolled clinical study is less than 12 weeks, or whose time since the last trial drug administration has not exceeded 5 half-lives (whichever is longer);
* Subjects positive for anti-drug antibodies against anti-epidermal growth factor receptor antibodies;
* Subjects with substance abuse, or who have used soft drugs within 3 months before screening or hard drugs within 1 year before screening; or who consume excessive tea, coffee, and/or caffeinated beverages daily (more than 8 cups, 1 cup = 250 mL); or who have a positive urine drug screen;
* Subjects with alcoholism, or whose weekly alcohol consumption exceeds 14 units within 3 months before screening (1 unit = 17.7 mL ethanol, i.e., 1 unit = 357 mL of beer with 5% alcohol content, 43 mL of liquor with 40% alcohol content, or 147 mL of wine with 12% alcohol content); or who have a positive alcohol breath test; and those who cannot cooperate with alcohol prohibition during the study;
* Subjects who smoked more than 10 cigarettes per day on average within 6 months before screening;
* Subjects who engaged in strenuous activities within 72 hours before drug administration, or cannot avoid strenuous activities during the study; or have other physiological or pathological conditions that may affect the absorption, distribution, metabolism, or excretion of the study drug;
* Subjects who have donated blood (including component blood) or lost more than 400 mL of blood, or received blood transfusions within 3 months before screening; or donated blood (including component blood) or lost more than 200 mL of blood within 1 month before screening;
* Subjects with a known history of allergy to the active ingredient or any excipient of the study drug, or to other biological products; or with a history of atopic allergic diseases (e.g., asthma, urticaria, eczematous dermatitis, etc.); or with allergic diathesis;
* Subjects who cannot tolerate venipuncture or have a history of fainting due to needle or blood;
* Subjects with special dietary requirements who cannot accept the diet provided by the clinical trial center;
* Subjects who cannot take effective contraceptive measures or plan to donate sperm within 3 months after the administration of the study drug;
* Other conditions deemed by the investigator to make the subject unsuitable for participating in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 86 (Estimated)
Dates: Start 2025-11-11 (Estimated); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞ | From enrollment to the end of treatment at 28 days
  Area under the concentration time curve extrapolated to infinity

SECONDARY OUTCOMES:
AUC0-t | From enrollment to the end of treatment at 28 days
  Area under the concentration time curve from time zero to the last measurable time point.
Cmax | From enrollment to the end of treatment at 28 days
  Peak concentration.
Tmax | From enrollment to the end of treatment at 28 days
  time to peak
t1/2 | From enrollment to the end of treatment at 28 days
  half-life
λz | From enrollment to the end of treatment at 28 days
  Terminal Elimination Rate Constant
CL | From enrollment to the end of treatment at 28 days
  clearance
Vd | From enrollment to the end of treatment at 28 days
  volume of distribution
Immunogenicity | From enrollment to the end of treatment at 28 days
  Anti-drug antibody positive rate
Adverse Event | From enrollment to the end of treatment at 6 months
  Incidence and Severity of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Jia, PhD, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
After the study result is published, email the application registration contact or the study leader to obtain it.